CLINICAL TRIAL: NCT01608087
Title: Pharmacokinetics and Safety of BI 695502 in Healthy Subjects: a Randomized, Single-blind, Single-dose, Parallel-arm, Active-comparator Clinical Phase I Study
Brief Title: Pharmacokinetics and Safety Study of BI 695502 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1302.1
Record Dates: First submitted 2012-05-22; First posted 2012-05-30 (Estimated); Results first posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Healthy
MeSH Terms: interventions — Bevacizumab

ARMS (3):
- BI 695502 (Experimental): Subject to receive one intravenous (i.v.) infusion of BI 695502
  Interventions: Drug: BI 695502
- bevacizumab A (Active Comparator): Subject to receive one i.v. infusion of bevacizumab
  Interventions: Drug: bevacizumab
- bevacizumab B (Active Comparator): Subject to receive one i.v. infusion of bevacizumab
  Interventions: Drug: bevacizumab

INTERVENTIONS:
Drug: BI 695502 — BI 695502 single i.v. infusion
  Arms: BI 695502
Drug: bevacizumab — bevacizumab single i.v. infusion
  Arms: bevacizumab B
Drug: bevacizumab — bevacizumab single i.v. infusion
  Arms: bevacizumab A

SUMMARY:
This trial will investigate the pharmacokinetics and safety of BI 695502 and to establish pharmacokinetic biosimilarity of BI 695502 compared to bevacizumab.

ELIGIBILITY:
Inclusion criteria:

1. Healthy males.
2. Complete medical history, including physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests.
3. Aged 21 to 50 years.
4. Body mass index below or equal to 30.
5. Body weight 65 to 95 kg, inclusive.

Exclusion criteria:

1. Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance.
2. Any evidence of a clinically relevant concomitant disease, as judged by the investigator.
3. History of relevant orthostatic hypotension, fainting spells, or blackouts.
4. Chronic or relevant acute infections.
5. History of relevant allergy/hypersensitivity (including allergy to the study medications or its excipients).
6. Intake of prescribed or over-the-counter drugs within less than 6 half-lives of the respective drug prior to study drug administration or during the trial.
7. Participation in another trial with a study medication within two months prior to administration or during the trial (six half-lives).
8. Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day).
9. Inability to refrain from smoking during days of confinement at the study center.
10. Current alcohol abuse as judged by the investigator.
11. Current drug abuse, as judged by the investigator.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2012-05-01 (Actual); Primary Completion 2012-11-01 (Actual); Study Completion 2012-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (2):
- New Zealand (2):
  - 1302.1.002 Boehringer Ingelheim Investigational Site, Auckland NZ
  - 1302.1.001 Boehringer Ingelheim Investigational Site, Christchurch

REFERENCES:
- [Derived] Hettema W, Wynne C, Lang B, Altendorfer M, Czeloth N, Lohmann R, Athalye S, Schliephake D. A randomized, single-blind, Phase I trial (INVICTAN-1) assessing the bioequivalence and safety of BI 695502, a bevacizumab biosimilar candidate, in healthy subjects. Expert Opin Investig Drugs. 2017 Aug;26(8):889-896. doi: 10.1080/13543784.2017.1347635. Epub 2017 Jul 12. PMID 28651442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, single-blind, single-dose, parallel-arm, active comparator, Phase I clinical trial. The trial was planned to be conducted in two stages and subjects were to be randomly allocated in each stage. Based on the interim analysis finalized on 18 February 2013, the trial was closed after Stage 1, and Stage 2 was not conducted.
Pre-assignment Details: Subjects were randomized in a 1:1:1 ratio to receive BI 695502, United States (US)-licensed Avastin® or European Union (EU)-approved Avastin®.
Groups:
- BI 695502 (T): Subjects were administered a single dose of 25 milligram per millilitre (mg/mL) BI 695502 concentrate for solution for infusion.
- United States (US)-Licensed Avastin® (R1): Subjects were administered a single dose of 25 milligram per millilitre (mg/mL) US-licensed Avastin® solution for intravenous infusion.
- European Union (EU)-Approved Avastin® (R2): Subjects were administered a single dose of 25 microgram per millilitre (mg/mL) EU-approved Avastin® concentrate for solution for infusion.
Period: Overall Study
Arm/Group | BI 695502 (T) | United States (US)-Licensed Avastin® (R1) | European Union (EU)-Approved Avastin® (R2)
Started | 30 | 30 | 31
Completed | 30 | 28 | 31
Not Completed | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other Reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set: All subjects who received at least one administration of trial medication were included in the safety evaluation.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695502 (T) | United States (US)-Licensed Avastin® (R1) | European Union (EU)-Approved Avastin® (R2) | Total
Number analyzed (Participants) | 30 | 30 | 31 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.8 (6.5) | 28.8 (8.1) | 26.6 (5.4) | 27.4 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 30 | 30 | 31 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 4 | 4 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 2 | 3 | 2 | 7
  Black or African American | 0 | 0 | 0 | 0
  White | 23 | 22 | 22 | 67
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞).
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) is presented as adjusted geometric mean (gMean) and geometric coefficient of variation (%) (gCV%). Adjustment were made for treatment effect and weight.
Time Frame: Pharmacokinetic samples were collected predose, just before the end of the infusion, 2, 4, and 8 hours after the start of the infusion
Population: Pharmacokinetic (PK) set: The PK set included all subjects in the treated set (subjects who received at least one administration of trial medication) who provided at least one evaluable observation of a PK endpoint and had no important protocol violations relevant to the evaluation of PK biosimilarity.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter
Arm/Group | BI 695502 (T) | United States (US)-Licensed Avastin® (R1) | European Union (EU)-Approved Avastin® (R2)
Number analyzed (Participants) | 30 | 30 | 30
microgram*hour/milliliter | 7013.010 (19.52) | 7261.119 (15.57) | 7649.491 (18.29)
Statistical Analysis 1: Comparison: BI 695502 (T) vs United States (US)-Licensed Avastin® (R1); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 96.58, 93.93% CI 2-sided [88.54 to 105.35] — (T/R1) * 100; Least squares estimates of log-transformed PK endpoint for T and R1 were back transformed to original scale to get adjusted point estimator and interval estimates for the ratio of the geometric means for treatments
Statistical Analysis 2: Comparison: BI 695502 (T) vs European Union (EU)-Approved Avastin® (R2); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 91.68, 93.93% CI 2-sided [83.50 to 100.65] — (T/R2) * 100; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: United States (US)-Licensed Avastin® (R1) vs European Union (EU)-Approved Avastin® (R2); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 94.92, 93.93% CI 2-sided [87.14 to 103.40] — (R1/R2) * 100; [other analysis details as in outcome 1, analysis 1]

2. Secondary Outcome: Area Under the Concentration-time Curve of the Analyte in Plasma Over the Time Interval From 0 to the Time of the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point is presented as adjusted geometric mean (gMean) and geometric coefficient of variation (%) (gCV%). Adjustment was made for treatment effect and weight.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour/milliliter
Arm/Group | BI 695502 (T) | United States (US)-Licensed Avastin® (R1) | European Union (EU)-Approved Avastin® (R2)
Number analyzed (Participants) | 30 | 30 | 30
microgram*hour/milliliter | 6570.047 (20.68) | 6639.315 (18.46) | 7167.313 (19.72)
Statistical Analysis 1: Comparison: BI 695502 (T) vs United States (US)-Licensed Avastin® (R1); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 98.96, 90% CI 2-sided [90.97 to 107.64] — (T/R1) * 100; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695502 (T) vs European Union (EU)-Approved Avastin® (R2); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 91.67, 90% CI 2-sided [84.02 to 100.01] — (T/R2) * 100; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: United States (US)-Licensed Avastin® (R1) vs European Union (EU)-Approved Avastin® (R2); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 92.63, 90% CI 2-sided [85.18 to 100.74] — (R1/R2) * 100; [other analysis details as in outcome 1, analysis 1]

3. Secondary Outcome: Maximum Measured Concentration of the Analyte in Plasma (Cmax)
Description: Maximum measured concentration of the analyte in plasma (Cmax) is presented as adjusted geometric mean (gMean) and geometric coefficient of variation (%) (gCV%). Adjustment was made for treatment effect and weight.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram/milliliter
Arm/Group | BI 695502 (T) | United States (US)-Licensed Avastin® (R1) | European Union (EU)-Approved Avastin® (R2)
Number analyzed (Participants) | 30 | 30 | 30
microgram/milliliter | 23.783 (16.11) | 23.425 (25.15) | 25.505 (15.18)
Statistical Analysis 1: Comparison: BI 695502 (T) vs United States (US)-Licensed Avastin® (R1); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 101.53, 90% CI 2-sided [92.74 to 111.14] — (T/R1) * 100; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: BI 695502 (T) vs European Union (EU)-Approved Avastin® (R2); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 93.25, 90% CI 2-sided [87.12 to 99.81] — (T/R2) * 100; [other analysis details as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: United States (US)-Licensed Avastin® (R1) vs European Union (EU)-Approved Avastin® (R2); Test type: Equivalence — Commonly applied acceptance range for bioequivalence/biosimilarity is 80% to 125%; ANOVA; Analysis of variance (ANOVA) model on the logarithmic scale including effects'treatment' and 'weight'; gMean ratio = 91.85, 90% CI 2-sided [83.91 to 100.54] — (R1/R2) * 100; Least square estimates of log-transformed PK endpoint for R1 and R2 were back transformed to original scale to get adjusted point estimator and interval estimates for the inter-subject ratio of the geometric means for treatments

ADVERSE EVENTS:
Time Frame: From first drug administration to end of trial; up to 99 days.
Description: Any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a subject in a clinical investigation who received a pharmaceutical product. The recorded Adverse Event may not have had a causal relationship with this treatment.
Groups:
- European Union (EU)-Approved Avastin® (R2): Subjects were administered a single dose of 25 microgram per millilitre(mg/mL) EU-approved Avastin® concentrate for solution for infusion.
Arm/Group | BI 695502 (T) | United States (US)-Licensed Avastin® (R1) | European Union (EU)-Approved Avastin® (R2)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 25/30 | 19/30 | 21/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695502 (T) (N=30) | United States (US)-Licensed Avastin® (R1) (N=30) | European Union (EU)-Approved Avastin® (R2) (N=31)
Upper respiratory tract infection (Infections and infestations) | 11 | 6 | 13
Respiratory tract infection (Infections and infestations) | 3 | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 1
Headache (Nervous system disorders) | 9 | 6 | 4
Dizziness (Nervous system disorders) | 3 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 2 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 3 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 2 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2013-01-11): https://cdn.clinicaltrials.gov/large-docs/87/NCT01608087/Prot_000.pdf
  • Statistical Analysis Plan (2012-12-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT01608087/SAP_001.pdf